CLINICAL TRIAL: NCT05794074
Title: Role of Xanthophylls in Visual Function
Acronym: Xanthovision
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: APHP220293
Record Dates: First submitted 2023-02-03; First posted 2023-03-31 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2023-01

CONDITIONS: Nutrition Deficiency (Xanth Deficiency) Due to A Particular Kind of Food
MeSH Terms: interventions — Xanthophylls

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- lutéine (Experimental): 10 mg/d lutéine
  Interventions: Dietary Supplement: luteine
- zeaxanthine (Experimental): 10 mg/d zéaxanthine
  Interventions: Dietary Supplement: zeaxanthine
- lutéine and zeaxanthine (Experimental): 10 mg/d lutéine + 2 mg/d zéaxanthine
  Interventions: Dietary Supplement: luteine and zeaxanthine
- placebo (Placebo Comparator): same excipient used in the other arms with a carmine red dye
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: luteine and zeaxanthine — luteine and zeaxanthine
  Arms: lutéine and zeaxanthine
Dietary Supplement: luteine — luteine
  Arms: lutéine
Dietary Supplement: zeaxanthine — zeaxanthine
  Arms: zeaxanthine
Dietary Supplement: Placebo — Placebo
  Arms: placebo

SUMMARY:
Ecy of lutein supplementation alone, or zeaxanthin supplementation alone, or a combination of both, compared to placebo, on the evolution of macular pigment density (MPOD) measured by fundus photography in XANTH-deficient patients receiving enteral nutrition.

DETAILED DESCRIPTION:
Lutein and zeaxanthin are plant pigments belonging to the carotenoid family, and more precisely to the subfamily of xanthophylls (XANTH), which are oxygenated carotenoids. These phytochemicals are not synthesised by humans and are almost always present in our diet. They are significantly absorbed and transported in our body. They are present in various organs, e.g. the eye and the skin. They accumulate in very high concentrations in the central area of the human retina. Because of this high accumulation, it has been hypothesised that they play one or more specific roles in the eye. This has been confirmed by several studies which have shown that XANTHs are involved in protecting the eye from damage by certain light rays (blue) and age-related macular degeneration. Other studies suggest that XANTH may improve glare tolerance and contrast sensitivity. They may also improve sensitivity to red and green colour discrimination. However, identifying the exact relationship between XANTH and visual function in XANTH supplementation is complicated by two main problems. Firstly, XANTH supplementation does not always increase MPOD (Macular Pigment Optical Density), which is an indicator of the concentration of XANTH in the macula, because there are poor responders to XANTH, i.e. subjects who absorb it very poorly and/or transport it very poorly to the retina. Secondly, MPOD seems to reach a maximum value and a plateau, and increasing the dose of XANTH, or the duration of supplementation, does not increase MPOD further. This is particularly the case in individuals who already have a high MPOD, close to the maximum value, before supplementation because they often consume XANTH-rich foods, and/or because they are strong responders to XANTH. Therefore, although studies suggest a specific role for XANTH in visual function, the problem of initially high MPOD in some individuals, coupled with MPOD saturation, has not allowed previous studies to provide definitive evidence on their role(s) in visual function.

ELIGIBILITY:
Inclusion Criteria:

* On exclusive enteral nutrition for at least 6 months
* Exclusive enteral nutrition that is intended to be continued for at least 6 more months.
* No XANTH supplementation in the last 6 months.
* Able to sit up to allow visual examinations to be performed
* Sufficient understanding to perform visual examinations, at the discretion of the physician
* Written consent signed by the patient or agreement of their carer, trusted person, relative, family for patients with cognitive impairment (assessed using an MMS test). A patient with an MMSE test result ≤ 24 will be considered as having cognitive disorders.

Exclusion Criteria:

* Current treatment with hydroxychloroquine or any other drug known to cause ocular toxicity
* Visually impaired patient: patient unable to read text (font size 11) at close range, with visual correction if the patient usually wears it
* Unoperated cataracts in both eyes
* Pregnant or breastfeeding woman
* Patient under legal protection: guardianship or curatorship
* Participation in other research in the same field of dietary supplementation, which may interfere with the results of this research.

Secondary exclusion criteria :

* Absence of XANTH (lutein and zeaxanthin) deficiency* in the blood sample taken at inclusion.
* Physical, ophthalmological or cognitive characteristics, evaluated at the Quinze-Vingt ophthalmological examination, which do not allow a reliable measurement of MPOD or of all the settings of visual function.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2023-04-01 (Estimated); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
evolution of MPOD Baseline Vs M6 | Baseline, month 6
  Changes in MPOD by fundus photography (blue light autofluorescence) from baseline to 6 months of supplementation (M6) with lutein or zeaxanthin, or a combination of both, vs placebo.

SECONDARY OUTCOMES:
Linkage between MPDO and visual settings | Baseline, Month 6
  evaluate the relation between MPOD and visual accuity/settings
Linkage between MPOD and blood and xanth blodd count | Baseline, Month 4 and Month 13(option)
  evaluate the relation between MPOD and Xanth blood count
Measurement of visual accuity and settings | Baseline, Month 4, Month 7, Month 13(option)
  Measurement of visual accuity and settings assessed in a standardised manner at the Quinze-Vingt by :
  * Retinal structure assessed by OCT and adaptive optics
  * Visual acuity
  * Central macular sensitivity measured by microperimetry
  * Colour vision, especially in blue
  * Contrast sensitivity
  * Glare sensitivity and dark adaptation.
  * SLO Imaging